CLINICAL TRIAL: NCT04517240
Title: A Study on Protein Losing Enteropathy In Systemic Lupus Erythematosus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, DRRAMADAN, resident doctor, Assiut University
Other Study IDs: systemic lupus enteropathy
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: SLE
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: endoscopy — upper and lower endoscopy and fecal calprotectin test
  Other Names: fecal calprotectin test

SUMMARY:
The aim of the current study is to investigate if there is GIT involvement in pt's with SLE particularly protein losing enteropathy also its prevalence among the studied cases and it's relation to disease activity .

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is an autoimmune disease in which the body's immune system mistakenly attacks healthy tissue in many parts of the body. Symptoms vary between people and may be mild to severe. Common symptoms include painful and swollen joints, fever, chest pain, hair loss, mouth ulcers, swollen lymph nodes, feeling tired, and a red rash which is most commonly on the face. Often there are periods of illness, called flares, and periods of remission during which there are few symptoms Virtually every system and organ can be affected by SLE. Gastrointestinal symptoms are common in SLE patients, and more than half of them are caused by adverse reactions to medications and viral or bacterial infections. Though not as common as lupus nephritis, SLE-related gastrointestinal involvement is clinically important because most cases can be life-threatening if not treated promptly. Lupus mesenteric vasculitis is the most common cause, followed by protein-losing enteropathy, intestinal pseudo-obstruction, acute pancreatitis and other rare complications such as celiac disease, inflammatory bowel diseases, etc. Protein-losing gastroenteropathy (PLGE)is a condition characterized by profound edema and severe hypoalbuminemia secondary to excessive loss of serum protein from the gastrointestinal tract, clinically indistinguishable from nephrotic syndrome.

Gastrointestinal loss of albumin is harder to investigate, as is its etiology. Consequently, in patients with hypoalbuminemia in which other possible etiologies have been excluded, protein-losing enteropathy must be considered and persistently investigated. The diagnosis of lupus-associated protein-losing enteropathy relies on characteristic clinical and laboratory features of SLE and on the exclusion of other possible causes of protein loss. Usually there are no findings suggestive of lymphatic leakage, such as steatorrhea, lymphocytopenia, and hypogammaglobulinemia; complement levels were low and serum cholesterol was high in about 70% of the reported cases . No antibodies were specifically associated with protein-losing enteropathy.Colonoscopy in (PLGE)showed mucosal thickening in 44% of patients, and the majority of patients (52%) revealed no abnormalities; on the other hand, intestinal histology either revealed mucosal edema, inflammatory cell infiltrate, lymphangiectasia, mucosal atrophy or vasculitis in 80% of patients.Intestinal biopsy should be done to exclude other diseases but does not help in defining the etiopathogenesis of the protein loss. Intestinal biopsies were normal in many cases, and others showed nonspecific findings including mononuclear infiltration, lymphangiectasia, vasculitis, deposits of C3 in capillary walls, and shortened villi. Generally there are no lesions of the epithelial surface.calprotectin protein is found in large quantities in neutrophil granulocytes, where it represents 5% of total proteins and 60% of cytoplasmic proteins.In the presence of inflammatory processes, calprotectin is released following granulation of neutrophil granulocytes. In the case of an inflammation of the intestine, calprotectin can be detected in feces. Fecal dosing is the only one that can provide direct indications on the location of inflammation, while the dosage in serum or plasma shows a state of inflammation that can be present anywhere in the body of the analyzed patient.

ELIGIBILITY:
Inclusion Criteria:

- all patients should fulfill ACR(1997)criteria for diagnosis of SLE newly diagnosed and not received immune suppressive regimens

Exclusion Criteria:

* Patients with acute gastroenteritis (fever, diarrhea and vomiting) . Patients with renal failure . Patients with heart failure. Patients with hepatic failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pt with systemic lupus with decreased protine in serum and don't have any other disease causing decrease protein
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
early diagnosis of protein losing enteropathy in SLE | baseline
  pt with sle have protein losing enteropathy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perednia DA, Curosh NA. Lupus-associated protein-losing enteropathy. Arch Intern Med. 1990 Sep;150(9):1806-10. PMID 2203319